CLINICAL TRIAL: NCT00005283
Title: Risk Factors For Asthma in Laboratory Animal Allergy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2004; R01HL030532 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To identify risk factors which predispose individuals to develop asthma and other manifestations of allergic disease on exposure to laboratory animals in the workplace.

DETAILED DESCRIPTION:
BACKGROUND:

In 1982, asthma and allergy to laboratory animals among persons who worked with the animals gained increased recognition as an occupational health problem affecting researchers, veterinarians, technicians, animal handlers, and others. At that time, more than 90,000 workers across the United States were at risk due to their exposure to lab animals in the more than 1,100 facilities registered by the United States Department of Agriculture. Several surveys of exposed workers indicated a prevalence rate of allergic symptoms due to laboratory animal allergy ranging from 19-30 percent in animal workers. Asthma was also a frequent disease among animal workers; these surveys indicated that as many as 13-14 percent of exposed workers had asthma.

The problem of laboratory animal allergy and asthma involved a vast industry that included medical and veterinary colleges, research institutes and universities, pharmaceutical manufacturers, commercial laboratory animal producers, and hospitals.

DESIGN NARRATIVE:

Recruitment for this longitudinal study began in November 1983 and ended in July 1987. The initial visit consisted of an extensive interview to identify and to exclude those individuals with laboratory animal allergy, asthma, and other manifestations of allergy and to obtain an occupational history. Venipuncture was used to obtain serum for IgE and IgG antibody assays. Pulmonary function tests, including a methacholine challenge, were administered. Psychosocial questionnaires were administered. Subjects were evaluated at six month intervals with skin tests, venipuncture, and methacholine challenge. The degree of exposure to animal allergens was quantitated by aeroallergen sampling of workplace and personal breathing zone air and by work diaries.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1983-07; Study Completion 1990-06 (Actual)

REFERENCES:
- [Background] Corn M, Koegel A, Hall T, Scott A, Newill C, Evans R: Characteristics of Airborne Particles Associated with Animal Allergy in Laboratory Workers. Ann Occup Hyg, 32:435-446 (Suppl 1), 1988
- [Background] Evans R III, Summers RJ, Newill CA: Allergic Reactions Caused by Exposure to Animals. In: Lichtenstein LM, Fauci AS (Eds), Current Therapy in Allergy, Immunology and Rheumatology - III. BC Decker Inc, Toronto, Philadelphia, p 5-7, 1988
- [Background] Eggleston PA, Newill CA, Ansari AA, Pustelnik A, Lou SR, Evans R 3rd, Marsh DG, Longbottom JL, Corn M. Task-related variation in airborne concentrations of laboratory animal allergens: studies with Rat n I. J Allergy Clin Immunol. 1989 Sep;84(3):347-52. doi: 10.1016/0091-6749(89)90419-3. PMID 2778241
- [Background] Eggleston PA, Kagey-Sobotka A, Proud D, Adkinson NF Jr, Lichtenstein LM. Disassociation of the release of histamine and arachidonic acid metabolites from osmotically activated basophils and human lung mast cells. Am Rev Respir Dis. 1990 Apr;141(4 Pt 1):960-4. doi: 10.1164/ajrccm/141.4_Pt_1.960. PMID 1691604
- [Background] Eggleston PA, Ansari AA, Ziemann B, Adkinson NF Jr, Corn M. Occupational challenge studies with laboratory workers allergic to rats. J Allergy Clin Immunol. 1990 Jul;86(1):63-72. doi: 10.1016/s0091-6749(05)80124-1. PMID 2196304
- [Background] Evans R III, Fortney S, Menkes H, Newill C, Cohens BH: Biological Indicators of Susceptibility. In: Green GM, Baker F (Eds), Work, Health and Productivity. Oxford University Press, 1991.
- [Background] Newill CA, Prenger VL, Fish JE, Evans R 3rd, Diamond EL, Wei Q, Eggleston PA. Risk factors for increased airway responsiveness to methacholine challenge among laboratory animal workers. Am Rev Respir Dis. 1992 Dec;146(6):1494-500. doi: 10.1164/ajrccm/146.6.1494. PMID 1456566
- [Background] Ziemann B, Corn M, Ansari AA, Eggleston P. The effectiveness of the Duo-Flo BioClean unit for controlling airborne antigen levels. Am Ind Hyg Assoc J. 1992 Feb;53(2):138-45. doi: 10.1080/15298669291359401. PMID 1543130
- [Background] Newill CA, Eggleston PA, Prenger VL, Fish JE, Diamond EL, Wei Q, Evans R 3rd. Prospective study of occupational asthma to laboratory animal allergens: stability of airway responsiveness to methacholine challenge for one year. J Allergy Clin Immunol. 1995 Mar;95(3):707-15. doi: 10.1016/s0091-6749(95)70176-1. PMID 7897154
- [Background] Eggleston PA, Ansari AA, Adkinson NF Jr, Wood RA. Environmental challenge studies in laboratory animal allergy. Effect of different airborne allergen concentrations. Am J Respir Crit Care Med. 1995 Mar;151(3 Pt 1):640-6. doi: 10.1164/ajrccm.151.3.7881650.